CLINICAL TRIAL: NCT07388693
Title: Feasibility of Integrating Olfactory Cues Into Virtual Reality Cue Exposure for Patients With Alcohol Dependence
Status: Not yet recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alva Lütt, Alva Lütt, Dr. med., Psychiatrische Universitätsklinik der Charité im St. Hedwig Krankenhaus, 10115 Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: EA1/269/24
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence, Virtual Reality Cue Exposure, Olfactory
MeSH Terms: conditions — Alcoholism; Anosmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: VR Cue-Exposure Including Olfactory Cues — Virtual Reality Cue Exposure (NCT05861843, NCT06333457)

SUMMARY:
Alcohol dependence (AD) is a prevalent and burdensome clinical condition with high relapse rates. A central risk factor for relapse is craving for alcohol, which can be evoked by both real-world and virtual cues in immersive Virtual Reality (VR). In addition to visual and auditory stimuli, olfactory cues are increasingly recognized as important for creating realistic, multisensory VR environments. However, no systematic investigation has yet examined how olfactory cues embedded in VR-based Cue Exposure (VR-CE) influence cue-elicited craving. As part of the OLFA-VR (Effects of Olfactory Stimuli in Virtual Reality Cue Exposure on Craving in Alcohol Dependence) research project, the present feasibility study aims to evaluate the feasibility, tolerability and acceptability of implementing olfactory cues into VR-CE.

In addition, this study not only examines the general feasibility of alcohol-related olfactory cues in VR-CE but also explores which specific alcohol-related olfactory cues prove to be feasible.

The investigators hypothesize that implementing olfactory cues into VR-CE will be feasible and tolerable for patients with AD, with no preventable serious side effects caused by VR-CE. The investigators also hypothesize that VR-CE will induce craving in most patients.

DETAILED DESCRIPTION:
Twenty patients with alcohol dependence (AD), treated in an inpatient or outpatient psychiatric clinic, will be included in the study. Participants will receive written and verbal information about the study and informed consent for participation will be obtained. A screening for eligibility will then be conducted. Sociodemographic data will be collected, and screening for harmful alcohol use (Alcohol Use Disorders Identification Test, AUDIT) and assessment of AD severity (Alcohol Dependence Scale, ADS) will be performed.

Participants will be exposed to two types of Virtual Reality (VR) scenarios combined with corresponding olfactory cues: a neutral VR scenario with neutral visual and olfactory cues (rose), and an alcohol-related VR scenario with alcohol-related visual and olfactory cues (beer, white wine, red wine, vodka, schnaps). The VR-CE protocol comprises one exposure to the neutral VR-CE followed by five alcohol-related VR-CEs. The five alcohol-related VR-CEs will be presented in a randomized order, each pairing a visual cue with the corresponding olfactory cue for a specific beverage.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65 years
* diagnosis of alcohol dependence according to ICD-10 (F10.2)
* history of alcohol craving
* able to provide written informed consent

Exclusion Criteria:

* hyposmia
* dependence on substances other than alcohol and nicotine
* current alcohol intoxication (randomly tested by measurement of breath alcohol concentration)
* unable to understand the study information, consent form or principles of the study
* abstinence for less than 7 days or ongoing consumption of alcohol
* severe neuropsychiatric disorder (e.g. schizophrenia spectrum disorders, bipolar affective disorder) or substantial cognitive impairment
* serious illnesses affecting brain or heart function that influence physiological study parameters
* acute suicidality (or acute endangerment of others)
* concurrent pharmacological treatment targeting AUD (e.g. benzodiazepines) or craving (e.g. acamprosate, disulfiram, naltrexone, nalmefene) and further medication significantly influencing heart rate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcohol dependence treated in inpatient or outpatient psychiatric clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Integrating Olfactory Cues Into Virtual Reality Cue Exposure | Day 1, after each Virtual Reality Cue Exposure (VR-CE): questions regarding olfactory cue identification, olfactory perception of intensity, realism and congruence Day 1, after completion of all VR-CEs and assessments: dropout
  Questions regarding olfactory cue identification, olfactory perception of intensity (1=imperceptible-7=intensely perceptible), realism (1=unrealistic-7=realistic) and congruence with visual cue (1=incongruous-7=congruous), higher scores reflect higher feasibility; dropout
Tolerability of Integrating Olfactory Cues Into Virtual Reality Cue Exposure | Day 1, before the start of the Virtual Reality Cue Exposures (VR-CE): SAM, PANAS, FMS, SSQ Day 1, after each VR-CE: questions regarding tolerability, SAM, FMS Day 1, after completion of all VR-CEs: SAM, PANAS, FMS, SSQ
  Questions regarding tolerability of the technology and olfactory stimuli (1=unpleasant-7=pleasant), higher scores reflect higher tolerability Emotional side effects: Self-Assessment Manikin (SAM; valence, arousal and dominance, range -8 to 8 in steps of 2; -8=happy/tense/submissive feeling, 0=neither happy/tense/submissive nor unhappy/calm/submissive, 8=unhappy/calm/submissive) and Positive and Negative Affect Schedule (PANAS; positive affect: range 10-50, higher score reflects higher levels of positive affect; negative affect: range 10-50, lower score reflects lower levels of negative affect) Physical side effects (cybersickness): Fast Motion Sickness Scale (FMS; range 0-20, higher score reflects higher levels of cybersickness) and Simulator Sickness Questionnaire (SSQ; total score, range 0-48, higher score reflects more sickness; nausea factor, 0-27 range, higher score reflects more nausea; oculomotor factor, range 0-21, higher score reflects more oculomotor problems)
Acceptability of Integrating Olfactory Cues Into Virtual Reality Cue Exposure | Day 1, after each VR-CE: question regarding technical functionality Day 1, after completion of all VR-CEs: UEQ, semi-structured interview
  Question regarding technical functionality User experience: User Experience Questionnaire (UEQ; pragmatic quality, hedonic quality and overall scale: range -3 to +3, -3=most negative, 0=neutral, +3=most positive answer) Semi-structured interview including overall impression, perceived usefulness of the integration of olfactory cues into Virtual Reality Cue Exposure (VR-CE), perceived willingness to use, open-ended feedback

SECONDARY OUTCOMES:
Assessment of Initial Clinical Efficacy of Integrating Olfactory Cues Into Virtual Reality Cue Exposure | Day 1, before the start of the Virtual Reality Cue Exposures (VR-CE), after each VR-CE and after completion of all VR-CEs: VAS Day 1, after completion of all VR-CE: Semi-structured interview
  Craving: Visual Analogue Scale (VAS; range 0-10, higher score represents higher levels of craving) Semi-structured interview including perceived craving

CONTACTS AND LOCATIONS:
Overall Officials: Alva Lütt, Dr. med., Principal Investigator — Psychiatrische Universitätsklinik der Charité im St. Hedwig Krankenhaus, 10115 Berlin, Germany; Stefan Gutwinski, Prof. Dr. med., Principal Investigator — Psychiatrische Universitätsklinik der Charité im St. Hedwig Krankenhaus, 10115 Berlin, Germany
Locations (1):
- Psychiatric University Hospital Charité at St. Hedwig Hospital, Berlin, State of Berlin, Germany